CLINICAL TRIAL: NCT04091386
Title: Observational Study Evaluating the Physical Activity in a Subset of Damoctocog Alfa Pegol Treated Hemophilia A Patients Who Are Enrolled in the HEM-POWR Study.
Brief Title: Study to Learn More About the Physical Activity Level of Patients Suffering From Hemophilia A Treated With Damoctocog Alfa Pegol (LIFE ACTIVE Study)
Acronym: LIFE-ACTIVE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20748
Record Dates: First submitted 2019-08-30; First posted 2019-09-16 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia A
Keywords: Physical activity; Coagulation factor VIII; Joint health
MeSH Terms: conditions — Hemophilia A; Motor Activity | interventions — Factor VIII

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia A patients: Patients with hemophilia A who are being treated with Damoctocog alfa pegol (Jivi, BAY94-9027) in routine medical practice and are enrolled in Bayer-sponsored study NCT03932201
  Interventions: Drug: Damoctocog alfa pegol (Jivi, BAY94-9027)

INTERVENTIONS:
Drug: Damoctocog alfa pegol (Jivi, BAY94-9027) — Intervention is given as part of routine medical practice

SUMMARY:
In this study researcher want to learn more about the change of physical activity of hemophilia A patients treated with damoctocog alfa pegol. Patients enrolled in this study will be wearing a small device measuring daily active time. Researcher will compare these physical activity data with patient's clinical data including bleeding events to gain information on how bleeding levels are related to the activity level of the patients.

The study aims to enroll about 80 patients who are at the same time also participating in the HEM-POWR study (NCT03932201) evaluating the effectiveness and safety of damoctocog alfa pegol.

DETAILED DESCRIPTION:
The primary objective is to evaluate the change in physical non-sedentary activity as measured by the ActiGraph CentrePoint Insight Watch (ActiGraph LLC, Pensacola, Florida) after 1, 2 and 3 years of treatment with damoctocog alfa pegol.

Secondary objectives are to determine the

* Change in intensity of physical activity,
* Association between physical activities and clinical outcomes / patient-reported outcome scores/ number of bleeds,
* Percentage of patients achieving WHO-recommended levels of activity
* Actual wear time.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the HEM-POWR study (NCT03932201)
* Naïve to damoctocog alfa pegol prior to enrollment to HEM-POWR study
* Prescribed for prophylaxis treatment for hemophilia with damoctocog alfa pegol
* Patient is willing to wear the provided device
* Signed informed consent/assent to participate in LIFE-ACTIVE: Observational study evaluating the physical activity in a subset of damoctocog alfa pegol treated Hemophilia A patients who are enrolled in the HEM-POWR study

Exclusion Criteria:

* Hypersensitivity to any material of activity monitor (e.g. steel, rubber)
* Time gap between enrollment to HEM-POWR study and enrollment to LIFE-ACTIVE study is greater than 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hemophilia A receiving damoctocog alfa pegol during Bayer-sponsored study NCT03932201
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Time of physical non-sedentary activity per week | 30 days at baseline
Time of physical non-sedentary activity per week | 30 days at year 1
Time of physical non-sedentary activity per week | 30 days at year 2
Time of physical non-sedentary activity per week | 30 days at year 3
Category of physical non-sedentary activity | 30 days at baseline
  The intensity of physical activity are: combined moderate to vigorous intensity, light intensity, moderate intensity, and vigorous intensity
Category of physical non-sedentary activity | 30 days at year 1
  The intensity of physical activity are: combined moderate to vigorous intensity, light intensity, moderate intensity, and vigorous intensity
Category of physical non-sedentary activity | 30 days at year 2
  The intensity of physical activity are: combined moderate to vigorous intensity, light intensity, moderate intensity, and vigorous intensity
Category of physical non-sedentary activity | 30 days at year 3
  The intensity of physical activity are: combined moderate to vigorous intensity, light intensity, moderate intensity, and vigorous intensity

SECONDARY OUTCOMES:
Time of physical activity per week by intensity | 30 days at each visit (baseline, year 1, 2 and 3)
  Intensity categories of physical activity are: combined moderate to vigorous intensity, light intensity, moderate intensity, and vigorous intensity
Time of physical activity per week by intensity stratified by sedentary and locomotion activity | 30 days at each visit (baseline, year 1, 2 and 3)
  Intensity categories of physical activity are: combined moderate to vigorous intensity, light intensity, moderate intensity, and vigorous intensity. Sedentary = yes/no; locomotion = yes/no
Association between physical activity time per week and annualized bleeding rate (ABR) | 30 days at each visit (baseline, year 1, 2 and 3)
  ABR from HEM-POWR study
Association between physical activity time per week and joint annualized bleeding rate (JABR) | 30 days at each visit (baseline, year 1, 2 and 3)
  JABR from HEM-POWR study
Association between physical activity time per week and hemophilia joint health score (HJHS) | 30 days at each visit (baseline, year 1, 2 and 3)
  HJHS from HEM-POWR study
Association between physical activity time per week and PRO-scores for treatment satisfaction | 30 days at each visit (baseline, year 1, 2 and 3)
  Patient reported outcome (PRO) scores from the Hemophilia Treatment Satisfaction Questionnaire for Adults collected in HEM-POWR study
Association between physical activity time per week and PRO-scores for health-related life quality | 30 days at each visit (baseline, year 1, 2 and 3)
  Patient reported outcome (PRO) scores from the Hemophilia Quality Life Measures for adults and Hemophilia Quality of Life short form for children questionnaires collected in HEM-POWR study
Association between physical activity time per week and PRO-scores for work productivity/ activity impairment | 30 days at each visit (baseline, year 1, 2 and 3)
  Patient reported outcome (PRO) scores from the Work Productivity and Activity Impairment Scale questionnaire collected in HEM-POWR study
Percentage of children (under 18) with ≥60 min per day of moderate to vigorous intensity physical activity | 30 days at each visit (baseline, year 1, 2 and 3)
Percentage of adults (age 18 to 64) with ≥150 min per week of moderate to vigorous intensity physical activity or with ≥75 min per week of vigorous intensity physical activity | 30 days at each visit (baseline, year 1, 2 and 3)
Repeated measure correlation between change in amount of non-sedentary physical activity time per week and change in annualized bleeding rate (ABR) | 30 days at each visit (baseline, year 1, 2 and 3)
  ABR from HEM-POWR study
Repeated measure correlation between change in amount of non-sedentary physical activity time per week and change in joint annualized bleeding rate (JABR) | 30 days at each visit (baseline, year 1, 2 and 3)
  JABR from HEM-POWR study
Actual wear time per week | 30 days at each visit (baseline, year 1, 2 and 3)
Percentage of actual wear time per week | 30 days at each visit (baseline, year 1, 2 and 3)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - Center for Comprehensive Care and Diagnosis of Inherited Blood Disorders, Orange, California
  - Tulane University, New Orleans, Louisiana
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, Canada
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Slovenia
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Taiwan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.